CLINICAL TRIAL: NCT00937001
Title: Investigating the Histopathological and Clinical Significance of Critical Illness Myopathy as a Cause of Debilitating ICU-Acquired Weakness
Brief Title: Critical Illness Myopathy as a Cause of Debilitating ICU-Acquired Weakness
Acronym: MUSIC Plus
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Wes Ely, Professor of Medicine, Vanderbilt University Medical Center
Organization: Vanderbilt University Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 081235
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Myopathy; Cognitive Impairment
Keywords: myopathy; respiratory failure; cognitive impairment; delirium
MeSH Terms: conditions — Muscular Diseases; Cognitive Dysfunction; Respiratory Insufficiency; Delirium | interventions — Biopsy; High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biopsy/Ultrasound (Experimental)
  Interventions: Procedure: Biopsy/Ultrasound

INTERVENTIONS:
Procedure: Biopsy/Ultrasound — obtain muscle biopsies at approximately 14 days of ICU, muscle ultrasound at 3-4 timepoints

SUMMARY:
ICU-acquired weakness represents a common and often devastating disease process which affects greater than 50% of critically ill patients. This pathogenesis of this acquired disease is multifactorial and results in variable severity, ranging from mild, transient to severe, permanent dysfunction of peripheral nerves in additional to muscle. In affected patients, weakness may persist for months to years after the acute phase of their illness, and has been implicated as a major contributor to decreased functional status and quality of life. Muscle ultrasound has been validated for assessment of muscle size as well as diagnosis of myopathic and neuropathic changes in patients with other known neuromuscular diseases. The use of muscle ultrasound or other imaging modalities for diagnosis or monitoring of ICU-acquired weakness has not been studied, although a single study using muscle ultrasound has shown significant change in muscle size in ICU patients receiving high dose corticosteroids and a prolonged course of paralytic agents. The investigators plan to use multiple modalities to examine skeletal muscle catabolism, function, and structure in patients during critical illness and recovery. The investigators will combine physical exam, hand grip dynamometry, electrophysiologic studies, serum biomarkers, muscle biopsies, and muscle ultrasound to assess a group of critically ill patients during their hospital stay. The investigators will obtain additional data, including neuropsychiatric assessments, severity of illness scores, administration of potentially harmful medications, and pertinent daily laboratory data. This study will last approximately 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be included if they are adult, patients in a medical and/or surgical ICU receiving treatment for any of the following:

* respiratory failure, or
* cardiogenic or septic shock.

Exclusion Criteria:

1. Cumulative ICU time > 5 days in the past 30 days, not including the current ICU stay, as this might create a state of flux regarding patients' cognitive baseline.
2. Severe cognitive or neurodegenerative diseases that prevent a patient from living independently at baseline, including mental illness requiring institutionalization, acquired or congenital mental retardation, known brain lesions, traumatic brain injury, cerebrovascular accidents with resultant moderate to severe cognitive deficits or ADL dependency, Parkinson's disease, Huntington's disease, severe Alzheimer's disease or dementia of any etiology.
3. ICU admission post cardiopulmonary resuscitation with suspected anoxic injury.
4. An active substance abuse or psychotic disorder, or a recent (within the past 6 months) serious suicidal gesture necessitating hospitalization. This exclusion will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact.
5. Blind, deaf, or unable to speak English, as these conditions would preclude our ability to perform the follow-up evaluation interviews.
6. Overly moribund and not expected to survive for an additional 24 hours and / or withdrawing life support to focus on comfort measures only.
7. Prisoners.
8. Patients who live further than 200 miles from Nashville and who do not regularly visit the Nashville area.
9. Patients who are homeless and have no secondary contact person available. This exclusion will enrich follow-up rates by avoiding patients with whom it is particularly challenging to maintain long-term contact.
10. The onset of the current episode of respiratory failure, cardiogenic shock, or septic shock was > 72 hours ago.
11. Patients who have had cardiac bypass surgery within the past 3 months (including the current hospitalization).
12. Patients with known Neuromuscular disease prior to admission.
13. BMI > 40 or patient size that will not make percutaneous muscle biopsy and muscle ultrasound possible.
14. Patients with a platelet count of less than 30,000.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2008-11; Primary Completion 2010-01 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To study the hypothesis that percutaneous muscle biopsy findings consistent with denervation atrophy and myopathic changes will correlate positively with the following assessments of peripheral muscle function. | 12 months

SECONDARY OUTCOMES:
To study the hypothesis that changes in size and density of pre-selected individual muscles, as assessed by serial bedside ultrasound, will correlate positively with the following assessments of muscle structure and function. | 12 months
To study the hypothesis that development of and duration of neurocognitive impairment during critical illness will correlate with changes in muscle size and appearance as measured by serial muscle ultrasound. | 12 months
To study the hypothesis that serum and muscle levels of pro-inflammatory cytokines, including IL-1, IL-6, TNF-alpha will correlate with development of ICU-Acquired weakness, as defined by characteristic muscle histopathologic findings or muscle loss. | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hooper, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- See also: ICU Delirium and Cognitive Impairment Study Group website — http://www.ICUdelirium.org